CLINICAL TRIAL: NCT06969703
Title: Azole Susceptibility and Resistance Mechanisms Surveys in Pathogenic Fungi by the China Antifungal Resistance Surveillance Trial (CARST)-Fungi (2023-2024)
Brief Title: Azole Susceptibility and Resistance Mechanisms Surveys in Pathogenic Fungi by the CARST-fungi (2023-2024)
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024Res301-001
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-12

CONDITIONS: Fungal Disease
Keywords: Azole susceptibility; pathogenic fungi; resistance mechanisms; Resistance Surveillance
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — All the fungal isolates from the sterile sites, including blood, ascitic fluid, pleural fluid, cerebrospinal fluid, and pus, bronchoalveolar lavage fluid (BALF), central venous catheter (CVC) tips, biliary tract fluid and tissues of patients with invasive yeast infections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The China Antifungal Resistance Surveillance Trial (CARST-fungi) study, which has been starting in July 2019, is a multi-center, prospective, observational, and laboratory-based study of pathogenic fungal isolates causing IFDs. All fungal isolates recovered from clinical samples will be collected. For each episode of fungal isolation, the information including the patient's age, gender, the ward location, the time of sample collection, and specimen type will be collected. All isolates will be sent to the Research Center for Medical Mycology, Beijing, China, for further study including species identification and azole susceptibility testing. Azole-resistant mechanisms will be elucidated by gene sequencing or expression level assay for resistance-related genes.

DETAILED DESCRIPTION:
Invasive fungal diseases (IFDs) are life-threatening diseases with considerable morbidity and mortality, primarily occurring in immunocompromised and critically ill hosts. Azoles represent the most widely prescribed antifungal class for IFDs. However, azole-resistance has become a growing problem worldwide. The major resistance mechanisms include mutations or overexpression of the drug target gene ERG11/cyp51, and overexpression of drug efflux pumps. Different resistance mechanisms vary by species and geographic distribution, and the underlying mechanisms in some species have not been well defined. A better understanding of antifungal resistance mechanisms will provide insights to reclaim those antifungal drugs as an option for empiric treatment of IFDs. Thus, comprehensive survey of azole susceptibility and resistance mechanisms of pathogenic fungi plays a significant role in understanding epidemiology and antifungal susceptibility such that to guide empirical therapy and aid antifungal stewardship efforts.

Since antifungal susceptibilities of pathogenic fungi are changing gradually year by year, the investigator put forward the following objectives and hypotheses of our survey:

Objectives

1. To survey azole-susceptibility status and evolutionary trend of pathogenic fungi isolated from tertiary hospitals in China
2. To elucidate the mechanisms and characteristics of azole-resistance in different pathogenic fungi

Hypotheses

(1) By comparing with CARST-fungi (2019-2020 and 2021-2022), evolution of antifungal susceptibilities in pathogenic fungi will be elucidated (2) Mechanisms and characteristics of azole-resistance will be revealed in various pathogenic fungi Our survey is a non-clinical, prospective, observational, and laboratory-based study; thus, it is not related to enrollment and inclusion of patients.

1. Clinical fungal isolates collection By the CARST-fungi study, all fungal isolates recovered from sterile sites, including blood, ascitic fluid, pleural fluid, cerebrospinal fluid, and pus, bronchoalveolar lavage fluid (BALF), central venous catheter (CVC) tips, biliary tract fluid and tissues of patients with invasive yeast infections, will be collected. Additionally, strains from considered colonizers such as urine, feces, sputum, and the genital tract will be also included. For each episode of isolation, the information including the patient's age, gender, the ward location (e.g., department of emergency, ICU), the time of sample collection, and the specimen type will be collected. About 300-350 clinical fungal isolates are expected to be collected. All the isolates will be sent to the Research Center for Medical Mycology, Beijing, China, for further study including species identification and antifungal susceptibility testing.
2. Fungal species identification All clinical fungal isolates will be identified to the species level. Six colonies from primary culture plates will be subcultured and identified by amplifying the sequences of the internal transcribed spacer (ITS) region and 28S ribosomal subunit (D1/D2) for yeast isolates, and ITS, beta-tubulin, calmodulin for moulds. Those sequences will be aligned by using CBS database.
3. Azole susceptibility testing Azole susceptibility testing will be performed according to the Clinical and Laboratory Standards Institute (CLSI) M27-A4 microbroth dilution method for yeasts and CLSI M38-A3 for moulds, and the tested drugs including fluconazole, itraconazole, voriconazole, posaconazole, and isavuconazole will be tested. In the same time, amphotericin B and echinocandins will be included for comparison. The interpretation of susceptibility will be performed by applying the updated species-specific clinical breakpoints (CBPs) according to CLSI M60 document. In the absence of CBPs, isolates will be defined as having a wild-type (WT) or a non-WT (NWT) drug susceptibility phenotype according to the epidemiological cutoff values (ECVs) as determined by the CLSI M59 document . Cross-resistance will be defined as resistance to at least two antifungals of the same drug class. Multi-resistance will be defined as resistance to at least two classes of antifungal drug.
4. Resistance-related genes amplification and sequencing Genomic DNA of azole-resistant or non-WT fungal strains will be extracted using the QIAamp DNA Mini Kit . Full open reading frame and promoter region of resistance-related genes including ERG11 (for Candida spp.), PDR1 (for C. glabrata), and cyp51A, cyp51B, hmg1 (for Aspergillus spp.) will be amplified and sequenced. At the same time, FKS genes of echinocandin-resistant isolates will also be sequenced. The amplified products will be sent to the BGI Company for sequencing and the sequences will be aligned with the reference strain by using the online tool of Clustal Omega.
5. Quantitative real-time reverse-transcription (RT)-PCR The expression level of drug target genes (ERG11 for Candida spp. and cyp51A, cyp51B for Aspergillus spp.) and drug efflux transporter genes (CDR1, CDR2, MDR1, SNQ2 for Candida spp. and cdr1B,abcC for Aspergillus spp.) will be assayed by the following method. Suspensions of azole-resistant or non-WT fungal isolates cells freshly prepared in YPD or SDB medium will be grown at 35 °C to reach the mid-exponential phase. Total RNA will be extracted by using the RNeasy Mini kit following the manufacturer's instructions. The RNA will then be treated with RNase-free DNase according to the manufacturer's recommendations. cDNA will be synthesized using an Advantage RT-for-PCR kit according to the manufacturer's instructions. RT-qPCR will be performed on an Applied Biosystems ViiA7 Real-Time PCR system using SYBR green reagent. Optimal thermal cycling conditions are consisted of a 10-min initial denaturation at 95°C, followed by 40 cycles of denaturation at 95°C for 15 s, and annealing/extension at 60°C for 10 s. The experiments will be carried out in triplicate for each data point. The cycle threshold (CT) value of the gene will be normalized to that of internal control ACT1 gene. Relative gene expression will be calculated as the fold change in expression of the isolates, compared to the mean expression values in drug-susceptible control strains.

This survey is non-clinical and no need of description for drug supply that given to patients here.

ELIGIBILITY:
Inclusion Criteria:

* fungal disease

Exclusion Criteria:

* non-fungal disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The individuals with fungal disease
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The type and spectrum of azole-resistance in the pathogenic fungi | By the end of Dec. 2025

CONTACTS AND LOCATIONS:
Overall Officials: Wei Liu, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
I will share the information of all the fungal isolates. But, I am not sure if I will be able to share the fungal isolates.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Bassetti M, Garnacho-Montero J, Calandra T, Kullberg B, Dimopoulos G, Azoulay E, Chakrabarti A, Kett D, Leon C, Ostrosky-Zeichner L, Sanguinetti M, Timsit JF, Richardson MD, Shorr A, Cornely OA. Intensive care medicine research agenda on invasive fungal infection in critically ill patients. Intensive Care Med. 2017 Sep;43(9):1225-1238. doi: 10.1007/s00134-017-4731-2. Epub 2017 Mar 2. PMID 28255613
- [Background] Pfaller MA, Woosley LN, Messer SA, Jones RN, Castanheira M. Significance of molecular identification and antifungal susceptibility of clinically significant yeasts and moulds in a global antifungal surveillance programme. Mycopathologia. 2012 Oct;174(4):259-71. doi: 10.1007/s11046-012-9551-x. Epub 2012 May 13. PMID 22580756